CLINICAL TRIAL: NCT06958484
Title: Iparomlimab and Tuvonralimab Injection (QL1706) Combined With Bevacizumab for Postoperative Adjuvant Therapy in Hepatocellular Carcinoma (HCC) With High Risk of Recurrence: A Multicenter, Open-Label, Single-Arm, Phase II Study
Brief Title: Iparomlimab and Tuvonralimab Injection (QL1706) Combined With Bevacizumab for Postoperative Adjuvant Therapy in Hepatocellular Carcinoma (HCC) With High Risk of Recurrence
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XYFY2025-KL117-01
Record Dates: First submitted 2025-04-21; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: HCC - Hepatocellular Carcinoma; Adjuvant Treatment
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Iparomlimab and Tuvonralimab Injection (QL1706) plus bevacizumab (Experimental)
  Interventions: Drug: Iparomlimab and Tuvonralimab Injection (QL1706) plus bevacizumab

INTERVENTIONS:
Drug: Iparomlimab and Tuvonralimab Injection (QL1706) plus bevacizumab — The patients with high-risk recurrence will be treated with Iparomlimab and Tuvonralimab Injection (QL1706) in combination with bevacizumab for postoperative adjuvant treatment .

SUMMARY:
Evaluation of the efficacy and safety of Iparomlimab and Tuvonralimab Injection (QL1706) in combination with bevacizumab for postoperative adjuvant treatment of HCC with high-risk recurrence risk

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in this study and sign the informed consent form;
2. Age 18-100 years old, male or female;
3. Hepatocellular carcinoma confirmed by histopathology, cytology or imaging;
4. CNLC PHASE I-II;
5. After surgical resection or local ablation, the intraoperative pathology shows that there is no residual resection margin, or R0 is confirmed by imaging within 4~8 weeks after surgery;
6. Have at least one high-risk recurrence factor:

(Definition of high-risk recurrence factors: Definition of high-risk recurrence factors: after radical surgery: presence of a single tumor >5 cm in diameter; Number of tumors>=3; concomitant vascular invasion (microvascular invasion or Vp1-2); Tumor grade III-IV; Post-ablation: 1. Single tumor >2cm but <= 5cm; 2. Multiple tumors: 2-4, all tumors <= 5 cm); 7. ECOG PS score: 0~1 points; 8. Child-Pugh Liver Function Rating: Grade A (< = 6 points) 9. Expected survival time >=12 months; 10. The laboratory test values within 3 days before the first dose meet the following requirements:

1. Routine blood test: (except for hemoglobin, no blood transfusion, no use of granulocyte colony-stimulating factor [G-CSF], no correction with medication within 2 weeks prior to screening):

   Absolute neutrophil count >=1.5×10^9/L; Platelets >=75×10^9/L; Hemoglobin >=90 g/L;
2. Biochemical examination:

   serum albumin >=30g/L; Serum total bilirubin < = 1.5×ULN; ALT and AST <= 3×ULN; Serum creatinine < = 1.5×ULN; or Cr clearance >50 mL/min
3. International normalized ratio (INR) < = 1.2 or prothrombin time (PT) outside the range of normal controls < = 2 seconds;
4. urine protein <2 (if urine protein >=2, 24-hour (h) urine protein quantification can be performed, and 24-hour urine protein quantification <1.0g can be enrolled); 11. If you have hepatitis B virus (HBV) infection, if HBsAg is positive, you need to test for HBV-DNA, and the HBV-DNA needs to be <2000 IU/mL (if the site only has a copy/mL testing unit, it must be < 104 copy/mL); For subjects with HBV-DNA>=2000 IU/mL, at least 1 week of antiviral therapy (only nucleosides such as entecavir, tenofovir disoproxil fumarate, and tenofovir alafenol tablets are allowed) prior to the first dose, and the viral copy number decreased by more than 10-fold (1 lg) compared to before the first dose. For patients with HBV infection, antiviral therapy is required throughout the study. Hepatitis C virus (HCV)-RNA positive subjects must be on antiviral therapy as per treatment guidelines; 12. Women of childbearing potential must have a negative pregnancy test (βHCG) before starting the first dose. Women of childbearing potential and men (sexually active with women of childbearing potential) must agree to contraception during treatment and within 6 months of the last dose.

Exclusion Criteria:

1. It is known that there are fibrotic plate HCC, sarcomatoid HCC or mixed-type cholangiocarcinoma and HCC;
2. There is evidence of residual, recurrent or metastatic disease;
3. History of hepatic encephalopathy;
4. Previous receipt of allogeneic stem cell or solid organ transplantation, or on the waiting list for liver transplantation;
5. Any treatment before HCC resection or ablation, including systemic treatment (including experimental drugs) and local treatment, such as TACE; and subjects who received more than one cycle of adjuvant TACE treatment after surgical resection;
6. Within 5 years before the first medication, there is a history of malignant tumors other than HCC, with negligible risk of metastasis or death (such as 5-year OS rate > 90%), such as fully treated cervical carcinoma in situ, non-melanoma skin cancer, localized prostate cancer, ductal carcinoma in situ, or stage I uterine cancer;
7. Co-infection with HBV and HCV, co-infection with HBV and delta hepatitis virus infection;
8. History of idiopathic pulmonary fibrosis, organizing pneumonia (such as obliterative bronchiolitis), drug-induced pneumonia or idiopathic pneumonia, or chest CT scan at screening shows evidence of active pneumonia;
9. Active tuberculosis;
10. History of autoimmune diseases or immunodeficiency diseases, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener's granulomatosis, Sjogren's syndrome, Guillain-Barré syndrome or multiple sclerosis;
11. Severe infection within 4 weeks before the first medication, including but not limited to hospitalization due to complications of infection, bacteremia or severe pneumonia;
12. Received oral or intravenous antibiotic treatment within 2 weeks before the first medication;
13. Use of non-steroidal anti-inflammatory drugs (NSAIDs) for daily treatment of chronic diseases;
14. Have bleeding predisposition or significant evidence of coagulation dysfunction (without anticoagulant treatment);
15. Currently or recently using aspirin or full-dose oral or intravenous anticoagulants;
16. Hemorrhage events due to untreated or incompletely treated esophageal and/or gastric varices within 6 months before the first medication;
17. Major vascular diseases (such as aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months before the first medication;
18. Inadequate control of arterial hypertension (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure >= 90 mmHg) (based on the average value of >= 2 measurements of BP readings), allowing the above parameters to be achieved through the use of antihypertensive treatment; previous occurrence of hypertensive crisis or hypertensive encephalopathy;
19. Significant uncontrolled or symptomatic hypercalcemia (ionized calcium > 1.5 mmol/L, calcium > 12 mg/dL, or corrected serum calcium > ULN) within 6 months before the first medication;
20. Within 3 months of having severe cardiovascular diseases (such as NYHA class II or above heart disease, myocardial infarction or cerebrovascular accident), unstable arrhythmias or unstable angina pectoris;
21. Clinically significant ascites;
22. Within 6 months before the first medication, having a history of intra-abdominal inflammation, including but not limited to peptic ulcer, diverticulitis or colitis;
23. Within 6 months before the first medication, having a history of abdominal or tracheoesophageal fistula, gastrointestinal perforation or intra-abdominal abscess;
24. Severe, non-healing or ruptured wounds, active ulcers or untreated fractures;
25. Performed hollow needle biopsy or other minor surgeries within 3 days before the first medication, excluding the placement of vascular access devices. 26. Within 4 weeks prior to the first administration of the drug, underwent major surgery, or was expected to undergo major surgery during the study period;

27. Had previously used systemic immunostimulants or immune checkpoint blockade therapy; 28. Was expected to receive systemic immunosuppressive drugs (including but not limited to glucocorticoids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor-α [TNF-α] preparations) within 2 weeks prior to the first administration of the drug, or was expected to receive systemic immunosuppressive drugs during the study treatment period; 29. Was vaccinated with live vaccines within 30 days prior to the first administration of the drug, or was expected to receive such vaccines during the treatment period or within 5 months after the last administration; 30. Was known to be allergic to any study drug or excipients; 31. Was contraindicated from using the investigational drug, or had any other diseases, metabolic disorders, physical examination findings, or clinical laboratory findings that might affect the interpretation of results or place the patient at a high risk of treatment complications; 32. Had other factors considered by the investigator as unsuitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
One-year recurrence-free survival rate | From enrollment to the end of treatment at 1 year

SECONDARY OUTCOMES:
Relapse-Free Survival at 6 months, RFS6 | From enrollment to the end of treatment at 6 months
Relapse-Free Survival, RFS | From enrollment to through study completion, an average of 1 year
Time To Relapse, TTR | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first,assessed up to 24 months

IPD SHARING:
Plan to Share IPD: No